CLINICAL TRIAL: NCT04976491
Title: Based on the Special Disease Management of Crohn's Disease Diet Studies --a Multicenter, Randomized, Controlled and Open Label Study
Brief Title: Based on the Special Disease Management of Crohn's Disease Diet Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-257
Record Dates: First submitted 2019-11-14; First posted 2021-07-26 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CD-C-Food group: During the first 3 months，participants received EEN；In the second 3months , CD-C-Food group received received CD-C-food .
  Interventions: Dietary Supplement: CD-C-Food
- EEN group: During the period, participants received EEN for 6 months.
  Interventions: Dietary Supplement: EEN

INTERVENTIONS:
Dietary Supplement: CD-C-Food — CD patients combined with the characteristics of Chinese diet, remove the refined food, and combined with food intolerance detection method to check the corresponding food
  Groups: CD-C-Food group
Dietary Supplement: EEN — EEN goup received EEN continuously for 6 moths
  Groups: EEN group

SUMMARY:
This project plans to develop a new diet therapy suitable for China -- CD-C-food, which is more in line with the common diet of Chinese patients' eating habits and economic conditions, and its expected therapeutic effect and influence on intestinal microorganism are similar to that of EEN. In order to explore the influence of intestinal microorganisms and their metabolites on the clinical remission effect and inflammatory response of patients with CD-C-Food, and to reveal the possible internal mechanism， a randomized control of adult subjects with a healthy CD-Chinese-food diet, treatment group of CD patients and animal model will be conducted by using intestinal microbiome, bacterial metabolite analysis, inflammatory factors detection and other technical means.

DETAILED DESCRIPTION:
Exclusive Enteral Nutrition (EEN) is the only established dietary treatment for children with CD.Changes in diet affect the amount of short-chain fatty acids and branched-chain fatty acids produced by changing the composition of intestinal flora, leading to changes in intestinal state.Through the long-term clinical observation of our team, most patients with CD can achieve stable remission by removing the processed food and screening the corresponding food by combining the characteristics of Chinese diet with the food intolerance detection method. So, what kind of diet is suitable for the treatment of CD patients in China? The CD-Treat program, replacing the Western diet with Chinese diet, so as to design an individualized program CD-Chinese-food (CD-C-food) that is consistent with the eating habits of Chinese patients with CD. By comparing the effects of this individualized diet with EEN on inducing and maintaining remission in CD patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients who are clinically diagnosed as stable CD; the diagnosis of CD has evidence of clinical manifestations and endoscopy, and was confirmed by histopathological report, referring to the consensus opinion on the diagnosis and treatment of inflammatory bowel disease in 2018. CDAI (Crohn's disease activity index)<150 points is regarded as clinical remission.
2. Have reading ability, can access the Internet, use mobile phone WeChat and use application (APP) software with the assistance of oneself or family members;

Exclusion Criteria:

1. Active patients (referring to CDAI greater than 150);
2. CD patients who currently need or expect surgical intervention during the study period.
3. CD patients with symptoms or signs of perforation such as abdominal abscess, intestinal fistula, etc.
4. Patients with complete intestinal obstruction or fibrous stenosis with pre-stenosis dilation that require surgery to relieve the obstruction.
5. CD patients with colorectal tumors. Those who have EN contraindications (active gastrointestinal bleeding, severe esophageal and gastric varices, intestinal obstruction, abdominal cavity syndrome, etc.).
6. Pregnancy and breastfeeding patients.
7. Severe hemodynamics, unstable vital signs, or the presence of rapid progression or end-stage disease, are expected to die during the course of the study.
8. Patients diagnosed with short bowel syndrome or with ileostomy or colostomy.
9. Patients with severe liver and kidney dysfunction, active infection, or other reasons (such as previous infliximab anaphylactic shock) cannot tolerate the treatment drugs used in this study.
10. The patient is allergic to known ingredients of enteral nutrition or has no previous EEN for 12 weeks.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The trial was carried out in 6 IBD center hospitals in China. The heads of IBD centers in all hospitals are members of the CCCF Academic Committee. A total of 200 IBD cases are planned to be enrolled in 6 centers.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Remission rate of patients Maintain difference in remission rate | 6 months
  Clinical remission rate（Crohn's Disease Activity Index<150)

SECONDARY OUTCOMES:
Quality of life scale for IBD (inflammatory bowel disease) patients | 6 months
  Total score is 145, the higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital Zhejiang University School of Medicine, Zhengzhou, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04976491/Prot_SAP_001.pdf